CLINICAL TRIAL: NCT02297711
Title: Total ExtraPeritoneal (TEP) Versus Open Minimal Suture Repair for Treatment of Sportsman's Hernia/Athletic Pubalgia: A Randomized Multi-center Trial.
Brief Title: TEP Versus Open Minimal Suture Repair for the Sportsman's Groin
Acronym: SPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R03430
Record Dates: First submitted 2014-09-25; First posted 2014-11-21 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Total ExtraPeritoneal (Experimental): Total ExtraPeritoneal (TEP) technique in general anesthesiacanal from behind
  Interventions: Procedure: Total ExtraPeritoneal
- Open minimal suture repair (Active Comparator): Open minimal repair (OMR) technique in local or spinal anesthesia
  Interventions: Procedure: Open minimal suture repair

INTERVENTIONS:
Procedure: Total ExtraPeritoneal — This is a keyhole operation which will use one small incision at the 'belly button' followed by two small incisions of approximately 5mm in diameter below the 'belly button' . A lightweight mesh is then placed over the inguinal ligament to reinforce the weakness. This approach is keyhole in nature with visualisation of the inguinal canal from behind - posteriorly.
  Arms: Total ExtraPeritoneal
Procedure: Open minimal suture repair — This is best described as open minimal repair and involves a small incision into the groin of the affected side. Once the inguinal canal is exposed the back wall is repaired using a simple suture to reinforce the weakness. This approach is open surgery in nature with visualisation of the inguinal canal from in front - anteriorly.
  Other Names: Open technique (OMR)
  Arms: Open minimal suture repair

SUMMARY:
Sportsman's hernia is defined as a weakness or disruption of the posterior wall of the inguinal canal. Open hernia repair with or without mesh or laparoscopic techniques with mesh have been advocated in the treatment of sportsman's hernia and associated athletic pubalgia. The results of the operative treatment from single centers are reported to be good to excellent in between 70 - 90% of patients with the most promising results reported using an open minimal repair (OMR) technique. There are no randomized trials comparing open versus laparoscopic techniques regarding time for recovery and relief of pain. The aim of this randomized study is to compare the effectiveness of OMR technique in local or spinal anesthesia to endoscopic Total ExtraPeritoneal (TEP) technique in general anesthesia for the treatment of Sportsman´s hernia/athletic pubalgia. The primary endpoint is patient being free from intractable groin pain during sports activity or daily work four weeks after surgery.

DETAILED DESCRIPTION:
The prevalence of chronic groin pain in athletes and physically active adults is between 5 and 10 % (1-3). The groin area is vulnerable in contact sports such as soccer, ice hockey, and rugby that require sudden muscle contraction around the hip and lower abdomen, repetitive kicking and side-to-side motion. Common causes for chronic groin pain in such sports include adductor tendonitis, musculus rectus abdominis tendopathy, osteitis pubis (edema on MRI scans at pubic symphysis) or disruption of the posterior wall of inguinal canal, which are all referred to as athletic pubalgia (1-3). No exact pathophysiological mechanism for pain has so far been identified in sportsman's hernia (posterior inguinal wall deficiency). A tear of the abdominal wall in posterior inguinal canal or conjoined tendon (tendinopathy), with or without bulging of a hernia, is suggested to be typical for a sportsman's hernia (4-6). The tissue damage is similar as in an incipient direct inguinal hernia with or without bulge. Diagnosis of a sportsman's hernia can only be set in patients having a typical history and having a suspected posterior inguinal wall deficiency on careful clinical examination. Magnetic resonance imaging (MRI) should be performed to exclude other injuries in the groin area. Sometimes also ultrasonography (US) would be added in the diagnostic work-up. Although presenting with similarly symptoms, the clinical entity of ''sportsman's hernia'' is exclusively distinct from athletic pubalgia (7), which includes a more wide range of groin injuries, such as adductor tendonitis and/or inflammation of the pubic symphysis (8,9).

Treatment of chronic groin pain is aimed toward its specific pathology (1-3). The first line of management includes rest, muscle strengthening and stretching exercises, physiotherapy, anti-inflammatory analgesics, as well as local anesthetic and/or corticosteroid injections. In resistant cases, operative treatment might be considered. Various operative approaches in athlete's pubalgia have been proposed depending on the suspected nature of injury. These operative approaches include open (5,10) and laparoscopic methods of hernia repair (11-12), tenotomies of muscle tendons close to the pubic bone (13,14), as well as release or neurectomies of nearby nerves (6-7). The results of operative treatment are good to excellent in 70 to 90% of patients (1-3). There is no evidence-based consensus available to guide surgeons for choosing between various operative treatments of sportsman's hernia/athletic pubalgia (1). Both conventional open and laparoscopic repairs produce good results, although the latter may allow the patient to an earlier return to full sports activity.

Open minimal repair (OMR) technique in local or spinal anesthesia seems to be a promising surgical approach in the treatment of posterior inguinal wall deficiency (10). Recent one-center analysis of this technique reported full freedom of pain in 91% four weeks after operation, full recovery to sports after 2 weeks and good patient's satisfaction in 100%. The laparoscopic techniques are reported to give an excellent outcome in 80-90% of patients. These methods are more expensive and need to be performed under general anesthesia. The studies are also heterogeneous concerning the use of different types of mesh and fixation techniques (11-12). Comparative studies between the OMR technique and laparoscopic treatment of sportsman's hernia/athletic pubalgia are lacking. The OMR technique is developed solely to strengthen the posterior inguinal wall weakness using non-absorbable sutures, but theoretically the TEP technique may heal a wider area in groin utilizing a 10x15 cm mesh placed in the preperitoneal space behind the pubic symphysis and posterior inguinal canal (11).

The aim of this randomized study is to compare the effectiveness of OMR technique in local or spinal anesthesia to TEP technique in general anesthesia for treatment of Sportsman´s hernia/athletic pubalgia with the primary endpoint; patients being totally free from groin pain during sports activity four weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* both males and females either professional or non-professional athletes or physically active adults
* age 18-50 years
* unilateral or bilateral complains (in bilateral pain both sides are to be operated and the randomization is on patient level and not hernia level)
* chronic dull, diffuse groin pain lasting > 6weeks
* history, physical examination and MRI indicating sportsman's hernia/athletic pubalgia
* pain above inguinal ligament in the deep inguinal ring, may radiate inner thigh, scrotum or pubic bone
* minor radiating pain can be at adductor origin or symphysis pubis
* grade I-II edema at pubic symphysis on MRI scan is allowed (can be secondary after groin disruption)

Exclusion Criteria:

* patients not willing to participate
* inguinal or femoral hernia
* MRI reveals other major pathology (bursitis, hip injury, stress fracture etc)
* isolated adductor tendonitis with groin pain below inguinal ligament
* femoro-acetabular impingement (FAI)
* isolated severe osteitis pubis (marked x-ray changes; grade III edema in MRI)
* former surgery to the actual groin
* allergy to polypropylene or other contra-indication to surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2014-12-03 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is number of patients having relief of pain during sports activity (VAS scores 0-20, range 0-100) at four weeks after surgery. | 4 weeks

SECONDARY OUTCOMES:
Secondary end-points are time to resume low-level training and full-level training/competing. | 1 year
One year follow-up of post-surgery complications | 1 year
Costs of surgery | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Aali Sheen, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Central Manchester University Hospitals NHS Foundation Trust, Manchester, Manchester (Manchester Borough), United Kingdom

REFERENCES:
- [Derived] Sheen AJ, Montgomery A, Simon T, Ilves I, Paajanen H. Randomized clinical trial of open suture repair versus totally extraperitoneal repair for treatment of sportsman's hernia. Br J Surg. 2019 Jun;106(7):837-844. doi: 10.1002/bjs.11226. PMID 31162653